CLINICAL TRIAL: NCT01529671
Title: An Investigator And Subject Blinded, Sponsor Open, Randomized, Placebo Controlled, Multiple Dose Study To Investigate The Safety, Toleration And Pharmacokinetics Of Multiple Oral Doses Of Pf-05089771 In Healthy Subjects And In Subjects With Osteoarthritis Of The Knee
Brief Title: A Safety And Tolerability Study Of PF-05089771 In Healthy Subjects And In Subjects With Otseoarthritis Of The Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B3291011
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — PF-05089771

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1: Experimental intervention: PF-05089771 or placebo (Experimental): Subjects will receive multiple doses of PF-05089771 or placebo twice daily to investigate the safety/tolerability and Pharmacokinetics (PK) of PF-05089771.
  Interventions: Drug: PF-05089771
- Cohort 2: Experimental intervention: PF-05089771 or placebo (Experimental): Subjects will receive multiple doses of PF-05089771 or placebo twice daily to investigate the safety/tolerability and PK of PF-05089771.
  Interventions: Drug: PF-05089771
- Cohort 3: Experimental intervention: PF-05089771 or placebo (Experimental): Subjects with osteoarthritis of the knee will receive multiple doses of PF-05089771 or placebo twice daily to investigate the safety/tolerability and Pharmacokinetic (PK) of PF-05089771.
  Interventions: Drug: PF-05089771
- Cohort 4: Experimental intervention: PF-05089771 or placebo (Experimental): Elderly Subjects will receive multiple doses of PF-05089771 or placebo twice daily to investigate the safety/tolerability and Pharmacokinetic (PK) of PF-05089771.
  Interventions: Drug: PF-05089771
- Cohort 5: Experimental intervention: PF-05089771 or placebo (Experimental): Subjects will receive multiple doses of PF-05089771 or placebo twice daily to investigate the safety/tolerability and PK of PF-05089771.
  Interventions: Drug: PF-05089771

INTERVENTIONS:
Drug: PF-05089771 — PF-05089771 will be dosed as a suspension twice daily (BID)
  Arms: Cohort 1: Experimental intervention: PF-05089771 or placebo
Drug: PF-05089771 — PF-05089771 will be dosed as a suspension twice daily (BID)
  Arms: Cohort 2: Experimental intervention: PF-05089771 or placebo
Drug: PF-05089771 — PF-05089771 will be dosed as a suspension twice daily (BID)
  Arms: Cohort 3: Experimental intervention: PF-05089771 or placebo
Drug: PF-05089771 — PF-05089771 will be dosed as a suspension twice daily (BID)
  Arms: Cohort 4: Experimental intervention: PF-05089771 or placebo
Drug: PF-05089771 — PF-05089771 will be dosed as a suspension BID
  Arms: Cohort 5: Experimental intervention: PF-05089771 or placebo

SUMMARY:
The purpose of the study is primarily to determine the safety and toleration and pharmacokinetics of PF-05089771 following escalating multiple doses lasting for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects or female subjects of non-child bearing potential between the ages of 18 and 55 years, inclusive.
* elderly cohort : healthy male and/or female subjects of 65 and 74 years,
* cohort 3: subjects with osteoarthritis of the knee: Male or female subjects not of child bearing potential between the ages of 18 and 75 years inclusive at the time of entering the study.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Treatment with an investigational drug within 60 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* 12-lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec at Screening. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the subject's eligibility.
* Use of prescription or non-prescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* As an exception, acetaminophen/paracetamol may be used at doses of ≤1 g/day. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
* Blood donation of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Unwilling or unable to comply with the Lifestyle guidelines described in this protocol.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

for cohort 3: Evidence of relapse or recurrence of clinically significant endocrine, metabolic, pulmonary, hepatic, osteo-mio-artricular, gastrointestinal, cardiovascular, renal, , psychiatric or neurological disease, or neurological disease less than 28 days prior to screening.

Symptomatic OA of the hip ipsilateral to index knee which the patient considers more painful than the knee. History of diseases other than OA that may involve the index knee in the last 12 months prior to screening, including but not limited to: inflammatory joint diseases (i.e rehumatoid arthritis and gout), calcium crystal diseases, bursitis, tendinitis, tumors and cysts, ligament injuries, bone fractures, post-infective pathologies; widespread chronic pain conditions (ie, fibromyalgia) and neuropathic disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of PF-05089771 | Days 1-16
Maximum concentration (Cmax) for PF-05089771 in plasma (measured in ng/mL) | Days 1, 4 and 14
Tmax = Time of maximum concentration of PF-05089771 in plasma (hr) | Days 1, 6 and 14
AUCtau= Area under the curve from the time of dosing to the next dose (ng.hr/mL) | Days 1, 6 and 14
Elimination half life (hr) = rate of elimination of PF-05089771 after the final dose | day 14 PK samples collected only for 48 hours

SECONDARY OUTCOMES:
AUCinf = Area under the curve from the time of dosing extrapolated to infinity (ng.hr/mL) | Days 14, over 48 hours of PK samples collection
Daily pain score throughout the treatment period using an 11-point Numeric Rating Scale (NRS). | Days 14, every day over 24 hours
Daily time to ascend and descend stairs. | Days 14, every day over 24 hours
Daily pain following stair climbing and descending | Days 14, every day over 24 hours
Daily time for self paced walk | Days 14, every day over 24 hours
Daily pain following self paced walk. | Days 14, every day over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3291011&StudyName=A%20Safety%20And%20Tolerability%20Study%20Of%20PF-05089771%20In%20Healthy%20Subjects%20And%20In%20Subjects%20With%20Otseoarthritis%20Of%20The%20Knee